CLINICAL TRIAL: NCT04280588
Title: Efficacy of Fingolimod in the Treatment of New Coronavirus Pneumonia (COVID-19)
Brief Title: Fingolimod in COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ning Wang, MD., PhD., Doctor, First Affiliated Hospital of Fujian Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRCTA, ECFAH of FMU [2020]027
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: Fingolimod 0.5 mg
- Control group (No Intervention)

INTERVENTIONS:
Drug: Fingolimod 0.5 mg — Each patient in the fingolimod treatment group was given 0.5 mg of fingolimod orally once daily, for three consecutive days
  Arms: Treatment group

SUMMARY:
Although immune-inflammatory treatment is not routinely recommended to be used for SARS-CoV-2 pneumonia, according to the pathological findings of pulmonary oedema and hyaline membrane formation, timely and appropriate use of immune modulator together with ventilator support should be considered for the severe patients to prevent ARDS development. The sphingosine-1-phosphate receptor regulators Fingolimod (FTY720) is an effective immunology modulator which has been widely used in multiple sclerosis.The aim of this study was to determine whether the efficacy of fingolimod for a novel coronavirus disease (COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* The patients who were diagnosed with the common type of NCP (including severe risk factors) and severe cases of new coronavirus pneumonia;
* Aged 18 to 85 years;
* Patients or authorized family members volunteered to participate in this study and signed informed consent.

Exclusion Criteria:

* Patients with any history of bradyarrhythmia or atrioventricular blocks
* Patients who are participating in other drug clinical trials;
* Pregnant or lactating women;
* ALT / AST> 5 ULN, neutrophils <0.5, platelets less than 50;
* Definite diagnosis of rheumatic immune-related diseases;
* Long-term oral anti-rejection or immunomodulatory drugs;
* Patients with active pulmonary tuberculosis, with definite bacterial and fungal infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-22 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
The change of pneumonia severity on X-ray images | 5 day after fingolimod treatment
  The lesion change on X-ray images from day 5 to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Wan-Jin Chen, Fuzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code